CLINICAL TRIAL: NCT00677664
Title: Effects of Glatiramer Acetate (Copaxone) in the Nerve Fiber Layer Thickness and Retinal Function in Diabetic Patients After Pan- Retinal Photocoagulation (PRP), a Double- Masked Randomized Clinical Trial.
Brief Title: Effects of Copaxone in the Retinal Function in Diabetic Patients After Panphotocoagulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Augusto Paranhos Jr, PHD, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COP 001
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; panretinal photocoagulation; copaxone; nerve fiber layer thickness; retinal function
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Glatiramer Acetate; Coat Protein Complex I; Mannitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Group which received Copaxone
  Interventions: Drug: Glatiramer acetate (Copaxone)
- B (Placebo Comparator): Group which received Mannitol
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Glatiramer acetate (Copaxone) — Drug was offered by subcutaneous administration one week prior and in the three sections of PRP, one per week.
  Other Names: Copaxone (Glatiramer acetate, COP, Copolymer-1)
  Arms: A
Drug: Mannitol — Drug was offered by subcutaneous administration one week prior and in the three sections of PRP, one per week.
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the effects of Copaxone injections in retinal function and integrity in diabetic patients who underwent pan-retinal photocoagulation.

DETAILED DESCRIPTION:
Purpose: to evaluate the neuroprotective effect of Copaxone (Glatiramer acetate) injections in the nerve fiber layer thickness and retinal function in diabetic patients who underwent panretinal photocoagulation (PRP).

Study Design: Double- Masked Randomized Clinical Trial. The follow up period estimated is 12 months after the last PRP section. Patients enrollment: Thirty patients with severe nonproliferative or early proliferative diabetic retinopathy and no previous laser treatment were enrolled. They were divided into two groups: "A" which received Copaxone or "B"which received mannitol (placebo) using a block randomization. Both drugs were offered by subcutaneous administration one week prior and in the three sections of PRP, one per week. All patients received and signed a written inform consent approved by the research ethics committee of UNIFESP.

Chronogram: All patients received a full ophthalmic examination (best-corrected Log-Mar visual acuity, slit lamp examination, applanation tonometry, fundus biomicroscopy and indirect fundus examination); functional examination (Humphrey 24-2 SITA STANDARD visual field, Electroretingrams and FDT C-20 strategy visual field) and anatomic examination (Color digital photography and fluorescein angiography (FAG), GDX- VCC, Optical Coherence Tomography (OCT) and Heidelberg Retinal Tomography (HRT) before PRP and 1st,3rd,6th months and 1 year after laser, or whenever needed for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Males or females; Females must be post-menopausal for 6 months and must have a negative pregnancy test (serum β-HCG) prior to study entry
* Age: 18 to 70 years old
* Type 1 or 2 diabetes, assigned for pan-retinal photocoagulation
* Vision acuity 20/100 or better
* SE of ±6,00 DE
* Volunteer must be willing and able to sign an informed consent
* Volunteer must be ambulatory and not requiring skilled nursing care
* Normal skin appearance in areas to be injected (no tattoo, scars, birth marks etc.)

Exclusion Criteria:

* Eye Related:

  * Dense cataract or vitreous opacity
  * Other retinal disease but diabetic retinopathy
  * Glaucoma (IOP higher than 21 mmHg and or Cup disk ratio equal higher than 0.8) or other optic nerve diseases
  * Other eye threatening systemic diseases
  * No ocular surgery in the last 6 months including laser treatment
  * No previous retinal photocoagulation or cryopexy of any kind
* Systemic exclusion criteria:

  * Known immunological condition/disease
  * No active infection within 30 days prior to enrollment (e.g. urinary tract infection, upper/lower respiratory tract infection, skin infection, arthritis etc.)
  * Use of interferons, immunosuppressive therapy, cytotoxic, corticosteroids, chemotherapy or lymphoid irradiation within 1 year prior to study entry.
  * Serious disease in the past or an unstable disease such as cancer, pulmonary, hepatic, renal, cardiovascular or metabolic diseases
  * History of alcoholism or drug addiction within the past year
  * Volunteer has participated in another clinical trial within the past 90 days or took an experimental drug within time scale of 5 x t1/2 of the experimental drug
  * Unstable psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-07; Primary Completion 2008-07 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Retinal function | one year

SECONDARY OUTCOMES:
Nerve fiber layer thickness | one year

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Paranhos Jr, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Perlman I, Gdal-On M, Miller B, Zonis S. Retinal function of the diabetic retina after argon laser photocoagulation assessed electroretinographically. Br J Ophthalmol. 1985 Apr;69(4):240-6. doi: 10.1136/bjo.69.4.240. PMID 4039601
- [Background] Stitt AW, Gardiner TA, Archer DB. Retinal and choroidal responses to panretinal photocoagulation: an ultrastructural perspective. Graefes Arch Clin Exp Ophthalmol. 1995 Nov;233(11):699-705. doi: 10.1007/BF00164672. PMID 8566826